CLINICAL TRIAL: NCT03203109
Title: Determinants of Balance Recovery After Stroke
Brief Title: Determinants of Balance Recovery After Stroke - Retrospective Study
Acronym: DOBRAS-R
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.126
Record Dates: First submitted 2017-05-02; First posted 2017-06-29 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Stroke
Keywords: lateropulsion; pusher syndrome; posture; balance; PASS; verticality perception; gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Postural Assessment Scale for Stroke (PASS) — Postural Assessment Scale for Stroke (PASS)

SUMMARY:
Retrospective cohort study of consecutive patients investigated in a neurorehabilitation ward after a first hemispheric stroke. Postural and gait disorders in relation to referential of verticality have been analyzed in routine care.

DETAILED DESCRIPTION:
300 consecutive patients, admitted in our department for neurorehabilitation after a first hemispherical stroke, have been enrolled retrospectively. During their hospitalisation, all patients have been routinely evaluated with clinical scales, evaluating motor and cognitive deficits. Postural and visual vertical (VV) assessments have been performed 1 to 4 times during in-patient-stay.

The objective was to analyse the determinants of balance recovery after stroke, in particular the impact of wrong referential of verticality.

Data collection was performed by means of medical records. Observation period covered from january 2012 to february 2018.

ELIGIBILITY:
Inclusion Criteria:

first hemispheric stroke patient non-opposed to inclusion

Exclusion Criteria:

history of neurological disorders interfering with balance history of vestibularly disorders interfering with balance unstable medical conditions history of cognitive disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients admitted in neurorehabilitation ward after first hemispheric stroke
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Posture | admission and monthly, up to 3 months
  Change from Baseline Score of Postural Assessment Scale for Stroke (PASS) at discharge

SECONDARY OUTCOMES:
Balance | admission and monthly, up to 3 months
  Assessment of Balance and Posture with SCP (Scale for Contraversive Pushing)
Gait | admission and monthly, up to 3 months
  Assessment of Gait with Lindmark test
Postural disorders | admission and monthly, up to 3 months
  Assessment of Postural control with CDP (Computerized posturography)
Visual vertical perception | admission and monthly, up to 3 months
  Assessment of the visual vertical (vv). Subject indicates which direction a visual line displayed on a computer screen (in darkness) is perceived as vertical in the roll plane.
Postural vertical perception | admission and monthly, up to 3 months
  Assessment of the postural vertical (pv). Subject is seated in a specific device (CE-marked) in darkness, and indicates which direction of her/his whole body is perceived as vertical in the roll plane.
Walking distance | admission and monthly, up to 3 months
  Assessment of walking distance with the 6-minute-walking-test (6-MWT)
Gait velocity | admission and monthly, up to 3 months
  Assessment of gait velocity at self-prefered-velocity on 10 meters
Pressure sensitivity (Hand and foot) | admission and monthly, up to 3 months
  Assessment of hypoesthesia with Semmes-Weinstein monofilaments test
Spasticity | admission and monthly, up to 3 months
  Assessment of Spasticity with Ashworth Scale
Laterality | admission and monthly, up to 3 months
  Assessment of Laterality with Edinburgh Handedness Inventory
Disability | admission and monthly, up to 3 months
  Assessment of Autonomy with FIM (Functional Independence Measure)
Neuropsychological Assessment 1 | admission and monthly, up to 3 months
  Assessment of Hemispatial Neglect with the Catherine Bergego Scale (CBS)
Neuropsychological Assessment 2 | admission and monthly, up to 3 months
  Assessment of Hemispatial Neglect with the fluff Test
Neuropsychological Assessment 3 | admission and monthly, up to 3 months
  Assessment of Hemispatial Neglect using 'thumb localizing test' (TLT)
Neuropsychological Assessment 4 | admission and monthly, up to 3 months
  Assessment of Hemispatial Neglect with the 'Comb and Razor Test'
Neuropsychological Assessment 5 | admission and monthly, up to 3 months
  Assessment of Hemispatial Neglect with the BEN ( Battery of tests for the quantitative assessment of unilateral neglect)
Neuropsychological Assessment 6 | admission and monthly, up to 3 months
  Assessment of Apraxia with ATS (Apraxia Screen of TULIA)
Neuropsychological Assessment 7 | admission and monthly, up to 3 months
  Assessment of Language with LAST (Language Screening Test)
Neuropsychological Assessment 8 | admission and monthly, up to 3 months
  Assessment of Aphasia with BDAE (Boston Diagnostic Aphasia Examination)
Neuropsychological Assessment 10 | admission and monthly, up to 3 months
  Assessment of depression with ADRS (Aphasia Depression Rating Scale)
Falls | at discharge, the number of falls is totalized
  Monitoring of falls occuring during the hospitalization
Visual field defect (hemianopia/quadranopia) | admission and monthly, up to 3 months
  standardized clinical examination
Identification of brain structures involved in the stroke | once, at 2 month
  anatomical MRI

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Pérennou, MD PhD, Principal Investigator — University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lafitte R, Diaine F, Dai S, Carre O, Dupierrix E, Jolly C, Piscicelli C, Perennou D. Writing and drawing tilts after right hemisphere stroke are signs of a wrong verticality representation. Ann Phys Rehabil Med. 2025 May;68(4):101923. doi: 10.1016/j.rehab.2024.101923. Epub 2025 Jan 15. PMID 39818122
- [Derived] Dai S, Piscicelli C, Marquer A, Lafitte R, Clarac E, Detante O, Perennou D. Improving orientation with respect to gravity enhances balance and gait recovery after stroke: DOBRAS cohort. Ann Phys Rehabil Med. 2024 Feb;67(1):101767. doi: 10.1016/j.rehab.2023.101767. Epub 2024 Jan 23. PMID 38266575
- [Derived] Perennou D, Chauvin A, Piscicelli C; Collaborators for the posturography study in the Determinants of Balance Recovery After Stroke (DOBRAS) cohort; Hugues A, Dai S. Determining an optimal posturography dataset to identify standing behaviors in the post-stroke subacute phase. Cross-sectional study. Ann Phys Rehabil Med. 2023 May;66(4):101707. doi: 10.1016/j.rehab.2022.101707. Epub 2023 Jan 4. PMID 36182062
- [Derived] Dai S, Piscicelli C, Clarac E, Baciu M, Hommel M, Perennou D. Lateropulsion After Hemispheric Stroke: A Form of Spatial Neglect Involving Graviception. Neurology. 2021 Apr 27;96(17):e2160-e2171. doi: 10.1212/WNL.0000000000011826. Epub 2021 Mar 15. PMID 33722996
- [Derived] Dai S, Piscicelli C, Lemaire C, Christiaens A, Schotten MT, Hommel M, Krainik A, Detante O, Perennou D. Recovery of balance and gait after stroke is deteriorated by confluent white matter hyperintensities: Cohort study. Ann Phys Rehabil Med. 2022 Jan;65(1):101488. doi: 10.1016/j.rehab.2021.101488. Epub 2021 Nov 11. PMID 33450367
- [Derived] Dai S, Piscicelli C, Clarac E, Baciu M, Hommel M, Perennou D. Balance, Lateropulsion, and Gait Disorders in Subacute Stroke. Neurology. 2021 Apr 27;96(17):e2147-e2159. doi: 10.1212/WNL.0000000000011152. Epub 2020 Nov 11. PMID 33177223